CLINICAL TRIAL: NCT04085003
Title: Nationwide Analysis of Intact Abdominal Aortic Aneurysm Repair in Portugal From 2000-2015
Brief Title: Intact Abdominal Aortic Aneurysm Repair in Portugal
Status: Completed | Type: Observational
Sponsor: Hospital Sao Joao (Other)
Responsible Party: Principal Investigator, Marina Felicidade Dias Neto, Principal Investigator, Hospital Sao Joao
Other Study IDs: NationwideAAAanalysis
Record Dates: First submitted 2019-09-08; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intact abdominal aortic aneurysm
  Interventions: Procedure: Endovascular repair or Open surgery
- Ruptured abdominal aortic aneurysm
  Interventions: Procedure: Endovascular repair or Open surgery

INTERVENTIONS:
Procedure: Endovascular repair or Open surgery — The outcomes of different types of repair will be obtained for intact and ruptured abdominal aortic aneurysm

SUMMARY:
Abdominal aortic aneurysm (AAA) repairs registered in the hospitals administrative database of the National Health Service from 2000 to 2015 were retrospectively analyzed regarding demographics (age and gender) and type of repair (open surgery [OS] or endovascular repair [EVAR]). Rate and mortality were compared among three time periods: 2000-2004, 2005-2009 and 2010-2015.

DETAILED DESCRIPTION:
All AAA interventions performed during the period 2000 to 2015 were retrospectively identified in a National Health Service (NHS) administrative database, the hospital morbidity database, formerly designated as Diagnosis-Related Groups (DRGs) database. This database was provided by the Portuguese Central Health System Administration (ACSS) and contains a registration of all hospitalizations (retrospective consecutive case entry) occurring in public hospitals in mainland Portugal.

Each episode includes information about diagnoses (primary and secondary diagnoses) and medical or surgical procedures, both coded using the International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9).

All admissions considered have a primary diagnosis ICD-9 codes for ruptured and non-ruptured AAA. The primary diagnosis of an episode represents the main condition investigated or treated during that hospital stay.

The rate of the repair was calculated based on the episodes of care with the above-mentioned disease ICD-9 codes plus the ICD-9 procedure codes suitable for AAA repair. Admissions with a primary diagnose of AAA that lacked a ICD-9 procedure code suitable for AAA repair were excluded, assuming that no repair was performed during that hospital stay. General indication for iAAA repair in Portugal are a maximum transverse diameter ≥5.5cm in men and ≥5.0 cm in women, as recommended by guidelines.

The number of deaths accounted for all patients that fail to be discharged alive from the hospital admission where the repair took place, irrespective to the direct cause of death. The number of admissions for repair in which the patient died divided by the number of all admissions for repair was used as a proxy of in-hospital mortality due to iAAA. The number of resident population in each year under analysis was provided by the National Institute of Statistics (INE) from 2000 to 2015. Resident population per year was used to calculate the rate of AAA repair and the death associated with AAA repair (thereafter mentioned as mortality to distinguish from the above-mentioned in-hospital mortality).

Death certificate with AAA-specific mortality was provided from the National Institute of Statistics (INE) from 2000 to 2015. INE data includes deaths outside the hospital besides those certificated at the hospitals.

In both databases, patients <50 years of age were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to abdominal aortic aneurysm repair in Portugal from 2000-20015

Exclusion Criteria:

* Patients without abdominal aortic aneurysm

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized in Portuguese public hospitals due to abdominal aortic aneurysm from 2000-2015.
  All patients that died in Portugal due to abdominal aortic aneurysm from 2000 to 2015.
Sampling Method: Non-Probability Sample
Enrollment: 6266 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of repair | longitudinal analysis from 2000 to 2015
  Number of repairs of abdominal aortic aneurysm in patients with more than 49 years old divided by the number of inhabitants above 49 years-old per year
Operative mortality | longitudinal analysis from 2000 to 2015
  Number of deaths after repair divided by the number or repairs per year

SECONDARY OUTCOMES:
Rate of mortality after repair | longitudinal analysis from 2000 to 2015
  Number of deaths after repair of abdominal aortic aneurysm in patients with more than 49 years old divided by the number of inhabitants above 49 years-old per year

IPD SHARING:
Plan to Share IPD: No